CLINICAL TRIAL: NCT05838950
Title: Detraining Effect of Short-term HIIT on Cardiometabolic Risk in Young Adults With Obesity
Brief Title: HIIT Effects on Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-010
Record Dates: First submitted 2023-02-13; First posted 2023-05-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Cardiovascular Diseases; Metabolic Disease; High-intensity Interval Training
Keywords: HIIT; Detraining effects; Cardiometabolic disease; Obesity; Young adults
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5s HIIT (Experimental): 5s HIIT group will perform one bout of sprint running for 5-seconds followed by 25-second, resting of total 40 repetition.
  Interventions: Other: high-intensity interval training intervention
- 10s HIIT (Experimental): 10s HIIT group will perform one bout of sprint running for 10-seconds followed by 50-second, resting of total 20 repetition.
  Interventions: Other: high-intensity interval training intervention
- 20s HIIT (Experimental): 20s HIIT group will perform one bout of sprint running for 20-seconds followed by 100-second, resting of total 10 repetition.
  Interventions: Other: high-intensity interval training intervention
- Control (Experimental): Control group
  Interventions: Other: high-intensity interval training intervention

INTERVENTIONS:
Other: high-intensity interval training intervention — Intervention groups include 3 arms with 3 different HIIT protocols to identify optimal exercise regimen for improving cardiometabolic health in young adults with obesity.

SUMMARY:
The primary aim of this randomized clinical trial is to compare the effects of three different HIIT protocols and a control group on cardiometabolic health in young adults with obesity. Participants will be randomly assigned to one of the following three groups, with each having varying work-to-rest ratios: 1) HIIT-A, 2) HIIT-B, 3) HIIT-C, and 4) control group. HIIT-A, HIIT-B, and HIIT-C groups will participate in six sessions of a running based HIIT program over a 2-week training period. Pre-clinical markers of cardiovascular disease, blood lipids and fasting glucose will be measured at the following three time points: baseline, post-intervention, and 2 weeks after the training cessation (i.e., measure for detraining effect). All measurements will be performed three days before the training program and three days after the intervention to avoid the effect of the last training session. Afterwards, the detraining test will be measured 2 weeks post intervention.

DETAILED DESCRIPTION:
Introduction: High-intensity interval training (HIIT) compared with other traditional exercise regimens has shown to be effective in improving cardiometabolic health (as measured by lipids, blood pressure [BP], insulin sensitivity, pulse wave velocity) in overweight and obese adults. By knowing which HIIT protocol is more efficacious in improving markers of cardiometabolic disease, exercise physiologists, researchers and clinicians can properly prescribe exercise medicine to obese young adults and possibly prevent disease progression. Therefore, the primary aim of the present research is to compare the effects of 3 different HIIT protocols compared with a control group on cardiometabolic health improvement in young adults with obesity.

Participants: Participants will be randomly assigned to one of the following three groups : 1) HIIT-A (5:25 s; 1:5 ratio), 2) HIIT-B (10:50 s; 1:5 ratio), 3) HIIT-C (20:100 s; 1:5 ratio), and 4) control group. HIIT-A, HIIT-B, and HIIT-C groups will participate in six sessions of running-based HIIT programs over a 2-week training period. The variables will be measured at the following three time points: baseline, post-intervention, and 2 weeks after the TC (i.e., measure for detraining effect).

High-Intensity Interval Training (six sessions over 2 weeks): Heart rate will be recorded - while performing a sprint running based on the wood court. The HIIT intensity will be set at 90% of the fastest baseline with 40 repetitions of 5-seconds work time, 20 repetitions of 10-seconds work time, or 10 repetitions of 20-seconds work time. All participants will perform one bout of sprint running for 5-, 10-, or 20- seconds followed by 25-second, 50-second, or 100-seconds resting. The supervisor will verbally encourage the running to inspire the sprint at "all-out" intensity. Note that a total of 200-seconds workout time is required per session.

ELIGIBILITY:
Inclusion Criteria:

* Young adults with obesity (Age 18 to 25 years old, BMI ≥ 30 kg/m2).

Exclusion Criteria:

* Syndromic obesity; 1) Any clinical symptoms including cognitive delay, 2) abnormalities in body structure(s), 3) organ-specific abnormalities (kidney, liver failure, excessive eating, and/or other signs of hypothalamic dysfunction such as fatigue, weakness and/or lack of interest in activities.
* Taking weight loss medication(s)
* Currently enrolled (or within previous 6 months) in a weight loss program;
* An underlying disease/medications (steroids, second generation psychotropic agents, hormonal contraception, statins, antihypertensive and antidiabetic medications) that could influence carbohydrate or lipid metabolism.
* Presence of cardiac pacemaker.
* Current or anticipated participation in another research that would interfere with any of the outcomes.
* Current or anticipated pregnancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Height | Baseline
  Height (cm)
Weight | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Weight (kg); Change from Baseline weight at 2 week and 4 week
Body mass index | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Body mass index (kg/m2); Change from Baseline BMI at 2 week and 4 week
Percentage body fat | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Percentage body fat (kg); Change from Baseline percentage body fat at 2 week and 4 week
Fat mass | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Fat mass (kg); Change from Baseline fat mass at 2 week and 4 week
Lean mass | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Lean mass (kg); Change from Baseline lean mass at 2 week and 4 week
Systolic blood pressure | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Systolic blood pressure (SBP, mmHg); Change from Baseline SBP at 2 week and 4 week
Diastolic blood pressure | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Diastolic blood pressure (DBP, mmHg); Change from Baseline DBP at 2 week and 4 week
Mean arterial pressure | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Mean blood pressure (MAP, mmHg); Change from Baseline MAP at 2 week and 4 week
Flow-mediated dilation | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Flow-mediated dilation (FMD, mm); Change from Baseline FMD at 2 week and 4 week
Carotid-femoral Pulse Wave Velocity (cPWV) | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  cPWV (m/s); Change from Baseline cPWV at 2 week and 4 week
Total cholesterol | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Total cholesterol (mg/dl); Change from Baseline TC at 2 week and 4 week
LDL-C | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  LDL-C (mg/dl); Change from Baseline LDL-C at 2 week and 4 week
HDL-C | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  HDL-C (mg/dl); Change from Baseline HDL-C at 2 week and 4 week
Triglycerides | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Triglycerides (TG, mg/dl); Change from Baseline TG at 2 week and 4 week
Glucose | Baseline, post test (2 weeks of intervention), training cessation (2 weeks of detraining)
  Glucose (mg/dl); Change from Baseline glucose at 2 week and 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Joon Young Kim, Ph.D, Principal Investigator — Syracuse University, Departments of Exercise Science
Locations (1):
- Women's Building, Syracuse, New York, United States